CLINICAL TRIAL: NCT06866288
Title: Belongingness in Nursing Through Mindfulness - BEING Mindful: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-036
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Mindfulness; Sense of Belonging
Keywords: Mindfulness based interventions; meditation; yoga; heart rate variability
MeSH Terms: interventions — Meditation; Yoga

STUDY DESIGN:
Intervention Model Description: Study Design This study is a minimal-risk, single-site, quasi-experimental study designed to evaluate the feasibility and preliminary efficacy of mindfulness-based interventions (MBIs) among faculty and staff at the University of New Mexico (UNM) College of Nursing (CON). Participants will be assigned to one of two intervention groups: (1) mindfulness meditation or (2) yoga. The study will assess psychosocial and physiological outcomes pre- and post-intervention.
  Blinding Blinding is not applicable in this study, as participants will be aware of their assigned intervention.
  Participant Selection and Eligibility Criteria Recruitment and Screening The study will use convenience sampling to recruit and enroll 60 participants from among the 71 faculty and 71 staff members at UNM CON. Study staff will contact interested individuals, who will undergo an eligibility screening via a one-page questionnaire (~5 minutes to complete). Screening will assess inclusion and exclusion criteria (Attac
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation (Experimental): Meditation is a practice of mental exercises designed to increase focus and cultivate a desire to relieve suffering in self and other. Many religious traditions have a form of meditation based practice. This study will focus on two forms of meditation both of which are focused on right mindfulness: 1) zazen which is a seated meditation primarily focused on the breath, posture, and sensation without attaching judgment. This is meant to develop awareness, equanimity, and insight, and 2) kinhin which is a walking meditation which is meant to connect mindfulness in one's movement by synchronizing breath and movement. It also focuses on development of awareness, equanimity, and insight. The two activities combined help the individual to nurture a thread of mindfulness. Instructors have developed a protocol to standardize the delivery of the meditation. Participants are requested to attend two meditation sessions per week.
  Interventions: Behavioral: Yoga
- Mindfulness Yoga (Active Comparator): Yoga is a holistic, multidimensional practice. There are three fundamental limbs of yoga: 1) breathwork (pranyanma), 2) physical postures with breathing techniques (asanas), and 3) meditation and visualization (Dhyana).) Yoga practice unites the mind, body and spirit leading to psychophysiological changes within the individual including improved self-regulation ability and stress response, mood, well-being, and quality of life. Yoga instructors will offer modifications and props such as blocks to ensure sessions are accessible to individuals of various abilities and minimize the risk of injury. Instructors have developed a detailed manual to standardize the delivery of the yoga intervention. Participants are requested to attend two yoga sessions per week.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — Each person will participate in seated meditation, then walking meditation, then return to seated meditation.
  Arms: Mindfulness Yoga
Behavioral: Yoga — Each person will participate in a yoga sessions.
  Arms: Mindfulness Meditation

SUMMARY:
The long-term goal of this study is to develop a mindfulness-based intervention (MBI) program to reduce stress and burnout while increasing belongingness and connectedness among faculty and staff at the University of New Mexico (UNM) College of Nursing (CON).

The central hypothesis is that the MBI intervention will improve psychosocial outcomes (sense of belonging) and physiological outcomes (heart rate variability, HRV) among CON faculty and staff. The specific aims are to:

Aim 1: Evaluate the feasibility and acceptability of MBIs (meditation or yoga) through participant interviews, recruitment, retention, and adherence rates.

Aim 2: Assess the preliminary effects of MBIs on psychosocial (burnout, stress, anxiety, sense of belonging) and physiological (HRV) outcomes. The hypothesis predicts improvements in both psychosocial and physiological measures post-intervention.

Researchers will compare meditation to yoga to see if one improves psychosocial and physiological outcomes better that the other.

Participants will be asked to:

* participate in meditation or yoga two times per week
* complete surveys
* use an app on their phone to answer short surveys
* wear a smart device

DETAILED DESCRIPTION:
Goal The primary goal of this study is to develop a mindfulness-based intervention (MBI) program aimed at reducing stress and burnout while enhancing a sense of belongingness and connectedness among faculty and staff at the University of New Mexico (UNM) College of Nursing (CON). This pilot project is an essential step toward achieving the long-term goal by evaluating the feasibility and preliminary efficacy of MBIs in an academic nursing environment.

Hypothesis and Specific Aims

The central hypothesis is that mindfulness-based interventions will lead to improvements in both psychosocial outcomes (such as sense of belonging, stress, anxiety, and burnout) and physiological outcomes (measured by heart rate variability, HRV) among CON faculty and staff. To assess this, the study aims to:

Aim 1: Evaluate the feasibility and acceptability of mindfulness interventions (meditation or yoga) for CON faculty and staff.

Feasibility will be determined by recruitment, retention, and adherence rates (percentage of training sessions attended).

Acceptability will be assessed qualitatively through participant interviews. Aim 2: Examine the preliminary effects of MBI (meditation or yoga) on psychosocial and physiological well-being.

Hypothesis 1: Psychosocial outcomes, including stress, burnout, anxiety, and sense of belonging, will improve after the intervention.

Hypothesis 2: Physiological outcomes, particularly HRV as measured through wearable devices, will show improvement post-intervention compared to pre-intervention.

Background and Significance Academic nursing faculty and staff play a crucial role in the preparation of future nurses. However, burnout, stress, and a lack of collegiality contribute to faculty shortages and hinder efforts to expand the nursing workforce. Studies have identified a strong connection between workplace stress and adverse behavioral, psychological, and physiological outcomes.

The 2024 American Association of Colleges of Nursing (AACN) Leading Across Multidimensional Perspectives (LAMP) Culture and Climate Survey emphasized the importance of belongingness for achieving academic nursing's mission. Despite existing strategies to foster belonging among students and faculty, there is a lack of clinical trials investigating interventions like mindfulness practices to enhance connectedness and well-being in nursing faculty and staff.

Mindfulness practices, including meditation and yoga, have been shown to improve mental health, interpersonal relationships, workplace communication, productivity, and resilience. Additionally, mindfulness is linked to improved autonomic nervous system (ANS) function and HRV, a key biomarker of stress and emotional regulation. This study addresses a significant research gap by evaluating the impact of MBIs on both psychosocial and physiological health markers in an academic nursing setting.

Preliminary Data

The UNM AACN LAMP Culture and Climate Survey (March-April 2023) assessed experiences of students, faculty, and staff at the College of Nursing. Faculty and staff responded to 10 items focused on belongingness, social connection, and feelings of isolation, revealing the following:

28% of faculty felt excluded during interactions at the CON. 30% of faculty felt their campus did not care about them. 39% of faculty felt isolated from others on campus. 38% of faculty lacked a sense of belonging within their academic community. 49% of faculty felt like a stranger when interacting with peers.

Faculty and staff suggested improving campus climate by:

Promoting a sense of belonging Building a stronger community Enhancing cohesiveness and collaboration These findings support the need for mindfulness-based interventions to improve faculty and staff well-being.

Scientific Rationale and Literature Support

Extensive research supports the benefits of mindfulness interventions:

Mindfulness reduces burnout and stress, improving workplace well-being. Yoga and meditation enhance emotional regulation and increase HRV, a physiological marker of stress resilience.

Workplace mindfulness practices improve communication, build shared goals, and enhance productivity while reducing employee turnover.

HRV is a well-established biomarker that reflects emotional and physiological regulation, making it a valid outcome measure for this study.

By integrating mindfulness interventions, this study aims to contribute valuable insights into strategies for improving faculty and staff wellness in academic nursing.

Study Design

The study is a minimal-risk, single-site, quasi-experimental design. Participants will be assigned to one of two MBI groups:

Mindfulness Meditation Group Yoga Group

Duration: The intervention will last six weeks, with participants attending regular in-person sessions.

Assessments:

Participants will complete pre- and post-intervention assessments to measure:

Psychosocial outcomes: Sense of belonging, burnout, stress, and anxiety. Physiological outcomes: HRV, assessed through wearable devices.

Study Population:

The UNM College of Nursing employs approximately 71 faculty and 71 staff. Using convenience sampling, 60 participants will be recruited (30 per group).

Screening Procedures:

Interested individuals will be contacted by study staff and screened for eligibility.

A short screening questionnaire (Attachment A) will assess inclusion/exclusion criteria.

Participants will also complete an Exercise Participation Screening (Attachment B) following the American College of Sports Medicine (ACSM) guidelines.

Outcome Measures:

Feasibility and acceptability (measured by recruitment, retention, adherence, and participant feedback).

Psychosocial health: Changes in stress, burnout, anxiety, and sense of belonging.

Physiological health: HRV improvements as measured by wearable devices.

Significance and Expected Impact:

Addresses a critical gap in nursing faculty and staff well-being research. Supports the AACN's recommendation to foster belongingness in academic nursing. Contributes to broader efforts in reducing burnout and improving workplace culture in nursing education.

Provides pilot data for future large-scale clinical trials on mindfulness in academic environments.

This study represents a crucial step in integrating mindfulness practices as a wellness strategy for nursing faculty and staff, with the potential to improve job satisfaction, retention, and overall mental and physical well-being.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* in general good health
* employed as College of Nursing (CON) faculty or CON staff
* reside in the state of New Mexico and able to attend 6 weeks of in-person research sessions
* willing to complete research assessments
* own a smart phone

Exclusion Criteria:

• major medical illness making individual unable to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Belongingness | Baseline and 6 weeks
  Belonging will be assessed using the 8-item Sense of Belonging Scale (SBS). The SBS measures the sense of belongingness or feelings of acceptance and inclusion in a community experienced by an individual.21 The SBS was developed to be adapted to specific contexts.21 Using the method described by Mellinger and Park (2023), we adapted the scale to be specific to UNM CON faculty and staff.
  Response categories range from 1 (Strongly disagree) to 5 (strongly agree). Responses are summed and the mean is calculated with higher scores corresponding to a stronger sense of belonging.22 The SBS-8 demonstrated high levels of reliability with a Cronbach's alpha coefficient of .96.21
Burnout | Baseline and 6 weeks
  Assessment of burnout: The Copenhagen Burnout Inventory is a valid and reliable, 19- item, self-report measure of burnout.24 Originally designed to measure burnout in among human service workers, it includes 3 scales. The personal burnout scale has six items and measures prolonged physical and emotional exhaustion. The work-related burnout scale has seven items that measure prolonged physical and emotional exhaustion secondary to work. The third scale, client-related burnout, has six items that measure burnout related to working with clients (client may be patients, students, service recipients). Each subscale can be scored separately.24 The three subscales have demonstrated good reliability and criterion related validity in a variety of samples.24,25

SECONDARY OUTCOMES:
Stress | Baseline and 6 weeks
  Stress will be assessed by the NIH toolbox measure of perceived stress; a 10-item fixed form. Responses are measured on a 5-point Likert scale ranging from 1 (Never) to 5 (Very Often) with higher scores indicating higher levels of perceived stress.(S. Cohen et al., 1983; Gershon et al., 2013)
Anxiety | Baseline and 6 weeks
  Anxiety will be assess using the Generalized Anxiety Disorder-7 screener (GAD-7), a 7-item self-report-measure of generalized anxiety disorder.(Simpson et al., 2014) Response categories range from 0 (Not at all) to 3 (Nearly every day). Responses are summed (range, 0 to 21) with higher scores corresponding to more severe levels of anxiety.
Trait Mindfulness | Baseline and 6 weeks
  Trait mindfulness will be assessed using the 15-item Mindfulness Attention Awareness Scale (MAAS).(Brown & Ryan, 2003) The MAAS was designed to assess core characteristics of mindfulness. The MAAS has demonstrated consistent reliability with Cronbach's alpha coefficients ranging from .80 to .90 in undergraduate, community, and nationally sampled adult populations.(Brown & Ryan, 2003)
State mindfulness | 6 weeks
  State mindfulness will be measured using the 5-item MAAS-State scale completed on the IlumiIvu mobile ecological momentary assessment app (mEMA app). The MAAS-State was designed to assess the expression of the core characteristic of mindfulness in real-time.(Brown & Ryan, 2003). Participants will be asked to complete three mEMA assessments per day (morning, afternoon, and evening). An alert will be programmed to be sent at pre-determined times to remind the participant to complete the
Heart Rate Variability (HRV) | 6 weeks
  Ambulatory assessment of physiological processes within the context of an individual's daily life will occur through use of a wearable wrist electronic sensor. This platform provides direct, real-time data which is sent from the wearable sensor to the mEMA app, by Bluetooth.HRV data will be collected via a Garmin Vivosmart5® device. This device has been shown to produce reliable heart rate data with the mean absolute percentage error below the designated acceptable 10% threshold. Each participant will receive training for use of the sensor and written instructions will be provided for future reference. Participants will wear the device on their non-dominant hand in their daily environment every day for six weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Ruyak, Principal Investigator — UNM HSC
Locations (1):
- University of New Mexico College of Nursing, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will make all unidentified information available for other researchers to use. We are in the process of determining the best platform to share information when it is entirely unidentified.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT06866288/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT06866288/ICF_001.pdf